CLINICAL TRIAL: NCT07345559
Title: Prospective, Randomized, Multicenter, Controlled Trial Assessing the Personalization of Mean Arterial Pressure in Adult Patients With Cardiogenic Shock
Brief Title: Personalisation of Mean Arterial Pressure in Adult Patients With Cardiogenic Shock
Acronym: CARDIOPAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/01; 2024-A00253-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-11-27; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic shock; Inotropes; vasopressors; Mean arterial pressure; Central Venous Pressure; Organ dysfunction; Mortality
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized MAP (Experimental)
  Interventions: Other: Personalized MAP
- Standard MAP (Active Comparator)
  Interventions: Other: Standard MAP

INTERVENTIONS:
Other: Personalized MAP — Patients receive blood pressure management targeting a personalized MAP ranging from 65 mmHg + CVP to 75 mmHg + CVP, without exceeding 90 mmHg.CVP is measured via a central venous catheter positioned in the superior vena cava. After 48 hours, if tissue perfusion is restored, the MAP target may be reduced to 65-70 mmHg.
  Arms: Personalized MAP
Other: Standard MAP — Patients receive blood pressure management aiming for a standard MAP target of 65-70 mmHg, according to international guidelines for cardiogenic shock management.
  Arms: Standard MAP

SUMMARY:
Cardiogenic shock is a life-threatening condition characterized by inadequate cardiac output, leading to organ hypoperfusion and high mortality. Maintaining mean arterial pressure (MAP) is crucial, but standard targets may be insufficient due to venous congestion. Central venous pressure (CVP) can help assess effective perfusion pressure. This study investigates whether a personalized MAP target adjusted by CVP improves organ function and survival compared to standard MAP management.

DETAILED DESCRIPTION:
Cardiogenic shock is a severe and life-threatening condition. Its prognosis remains very poor with a high mortality rate (up to 50% in clinical series) despite recent therapeutic advances. Current recommendations suggest the use of inotropes and vasopressors to maintain tissue perfusion and prevent organ failure.

During cardiogenic shock, the mean arterial pressure (MAP) level is associated with survival. A post hoc analysis of a recent randomized trial found increased mortality among patients in cardiogenic shock whose average MAP was <70 mmHg during the first 36 hours after randomization, compared to patients with MAP ≥70 mmHg (58% vs. 29%, p<0.01). Another observational study found higher mortality among patients with a mean MAP <65 mmHg during the first 24 hours of shock compared to those with MAP ≥65 mmHg (57% vs. 28%, p<0.001). In this study, the incidence of renal failure was also inversely associated with MAP level. The optimal MAP target remains unknown during cardiogenic shock.

Due to the characteristic venous congestion, the effective perfusion pressure may be very low during cardiogenic shock despite MAP being within the usual target (65 mmHg). Furthermore, increased central venous pressure (CVP) is associated with higher mortality during cardiogenic shock. Considering venous congestion by measuring or estimating CVP is necessary to assess the effective perfusion pressure (MAP minus CVP) in order to protect against organ dysfunction. In this perspective, the MAP target should be increased by the value of the CVP.

The investigators hypothesize that personalizing the MAP target (to achieve an effective perfusion pressure of 65 mmHg) improves organ perfusion and survival during cardiogenic shock compared to the usual MAP target of 65 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Cardiogenic shock state, according to the consensus definition,
* SCAI (Society for Cardiovascular Angiography and Interventions) classification ≥ C
* Consent from the patient or close relative / trusted person or emergency inclusion procedure
* Benefiting fromciary of a social security scheme

Exclusion Criteria:

* Catecholamine infusion for more than 24 consecutive hours;
* CVP < 5 mm Hg at inclusion;
* MAP > 70 mmHg at inclusion;
* Chronic kidney disease stage G4 (defined by an eGFR between 15-29 ml/min/1.73 m²) or G5 (defined by an eGFR less than 15 ml/min/1.73 m²) according to the KDIGO CKD classification at inclusion;
* Chronic dialysis or presence of renal replacement therapy criteria at inclusion ;
* Recovered cardiopulmonary arrest within 7 days prior to inclusion;
* Patient already on mechanical circulatory support at inclusion before enrollment (patients who receive support after inclusion will not be excluded);
* Primary diagnosis of tamponade, pulmonary embolism, or septic shock;
* Hypersensitivity to norepinephrine tartrate or to any of the following excipients: sodium chloride, hydrochloric acid or sodium hydroxide water for injectable preparations;
* Absence of central venous access;
* Known pregnancy or current breastfeeding;
* Under legal guardianship, curatorship, or judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be a composite of mortality, use of cardiac mechanical circulatory support, and severe renal failure. | 7 days and 28 days after randomization

SECONDARY OUTCOMES:
Mortality in the intensive care unit (ICU), and in hospital | 28 days and 90 days after randomization
Length of stay in the ICU and in the hospital | 28 days and 90 days after randomization
Proportion of patients requiring cardiac mechanical circulatory support | 28 days after randomization
Proportion of patients requiring renal replacement therapy | 28 days after randomization
Proportion of patients with severe acute kidney injury (stage 2 and stage 3 according to KDIGO AKI classification) | 7 days after randomization
  Defined as stage 2 or stage 3 according to the Kidney Disease: Improving Global Outcomes (KDIGO) Acute Kidney Injury classification
Duration of inotrope and vasopressor support | 28 days after randomization
Use of mechanical ventilation | 28 days after randomization
Number of ventilator-free days | 28 days after randomization
Evolution of the vasoactive inotropic score (VIS) | 5 days after randomization
  The clinical outcome is defined based on the Vasoactive Inotropic Score (VIS), according to published standard references
Evolution of lactate levels | 5 days after randomization
Evaluation of mottling score | 5 days after randomisation
Evaluation of capillary refill time | 5 days after randomization
Evaluation of Sequential Organ Failure Assessment (SOFA) score | 5 days after randomization
  The clinical outcome is defined based on the Sequential Organ Failure Assessment (SOFA) score, according to published standard references
Proportion of patients with sustained ventricular and/or supraventricular arrhythmias | 5 days after randomization
Proportion of patients with stroke, non-cerebral ischemia, new or recurrent myocardial infarction | 28 days after randomization
Proportion of patients with major bleeding, defined according to the ISTH classification | 28 days after randomization
  Defined according to the International Society on Thrombosis and Haemostasis (ISTH) classification.
Net clinical benefit at D28 (survival without thrombotic event or major bleeding). | 28 days after randomization
Proportion of patients receiving new specific treatments after randomization during hospital stay | 28 days after randomization

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'Amiens-Picardie, Amiens
  - Hôpital Henri Mondor, Créteil
  - Hôpital Privé Jacques Cartier, Massy
  - CMC Ambroise Paré - Hartmann, Neuilly-sur-Seine
  - CHU d'Orléans, Orléans
  - Hôpital Lariboisière, Paris
  - Hôpital Cochin, Paris
  - Clinique NCT + /Saint-Gatien, Saint-Cyr-sur-Loire
  - Centre Cardiologique du Nord, Saint-Denis
  - CHRU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No